CLINICAL TRIAL: NCT04499339
Title: A Phase I/IIa Clinical Trial to Assess Feasibility, Safety and Antitumor Activity of Autologous SLAMF7 CAR-T Cells in Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CARAMBA-1; 2019-001264-30 (EudraCT Number)
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: SLAMF7; Chimeric antigen receptor; CAR; CAR-T cell; immunotherapy; virus-free gene transfer
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All eligible patients (Experimental)
  Interventions: Drug: SLAMF7 CAR-T

INTERVENTIONS:
Drug: SLAMF7 CAR-T — Single infusion of autologous SLAMF7 CAR-T cells

SUMMARY:
Multiple myeloma (MM) is a rare hematologic malignancy of aberrant plasma cells.

There is a high and currently unmet medical need for novel, innovative treatment concepts to improve the therapeutic outcome and prognosis of patients suffering from MM.

There is definitive evidence that MM is susceptible to immune-based therapies from pre-clinical investigations and early clinical trials.

CARAMBA-1 is a first-in-human clinical trial of adoptive immunotherapy with autologous signaling lymphocytic activation molecule F7 (SLAMF7) chimeric antigen receptor (CAR)-T cells in patients with advanced MM that have exhausted conventional therapies.

The CARAMBA-1 clinical trial is an open-label, non-randomized, multicenter clinical trial which combines a phase I dose-escalation part with a phase IIa dose-expansion part to assess feasibility, safety and anti-myeloma activity of SLAMF7 CAR-T cells.

The CARAMBA project and the CARAMBA-1 clinical trial are supported by the European Union in the Horizon 2020 research and innovation program.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a rare hematologic malignancy of aberrant plasma cells.

There is a high and currently unmet medical need for novel, innovative treatment concepts to improve the therapeutic outcome and prognosis of patients suffering from MM.

There is definitive evidence that MM is susceptible to immune-based therapies from pre-clinical investigations and early clinical trials.

CARAMBA-1 is a first-in human clinical trial of adoptive immunotherapy with autologous SLAMF7 CAR-T cells in patients with advanced MM that have exhausted conventional therapies.

The CARAMBA-1 clinical trial is an open-label, non-randomized, multicenter clinical trial which combines a phase I dose-escalation part with a phase IIa dose-expansion part to assess feasibility, safety and anti-myeloma activity of SLAMF7 CAR-T cells.

SLAMF7 CAR-T cells are manufactured using virus-free gene-transfer using the Sleeping Beauty transposon system.

The CAR-T cell product is formulated to contain equal proportions of CD8 cytotoxic and CD4 helper SLAMF7 CAR-T cells.

The CARAMBA project and the CARAMBA-1 clinical trial are supported by the European Union in the Horizon 2020 research and innovation program.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Patient is ≥18 years of age.
3. Patient is willing and able to adhere to the protocol requirements.
4. Patient with diagnosis of MM who has been treated with at least 2 prior lines of treatment, including at least one cycle of high-dose chemotherapy with autologous hematopoietic stem cell transplantation if the patient was eligible, and exposure to an immunomodulatory imide drug (e.g. lenalidomide and/or pomalidomide), a proteasome inhibitor, and an anti-CD38 antibody.

   (Note: Induction therapy, up to 2 cycles of high-dose chemotherapy with autologous hematopoietic stem cell transplantation, and subsequent consolidation and/or maintenance therapy are considered one line of treatment).
5. At least one of the following subcriteria must be measured in the patient:

   * Serum M-protein greater or equal to 0.5 g/dL
   * Urine M-protein greater or equal to 200 mg/24 h
   * Serum free light chain (FLC) assay: involved FLC level greater or equal to 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal
   * A biopsy-proven evaluable plasmacytoma
   * Bone marrow plasma cells >10% of total bone marrow cells (>30% if bone marrow plasma cells are the only marker of measurable disease)
6. Patients previously treated with an anti-SLAMF7 antibody are eligible.
7. Karnofsky performance status ≥60%. If patient has a Karnofsky performance status <60% (e.g. after a spinal cord injury) but is judged to be medically fit by the investigator, patient is eligible.
8. Female patients of childbearing potential must:

   1. have a negative pregnancy test (blood) at screening.
   2. either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective measures of contraception without interruption, from screening through 1 year following the investigantional medicinal product (IMP) infusion. A highly effective method of contraception or birth control (failure rate less than 1% per year when used consistently and correctly) must be practiced. The patient should be informed of the potential risks associated with becoming pregnant while enrolled in this clinical trial. Reliable methods for this trial are: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, sexual abstinence or vasectomized sexual partner. Abstinence is only accepted as true abstinence: when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods and withdrawal] are not acceptable methods of contraception.) Postmenopausal (no menses for at least 1 year without alternative medical cause) or surgically sterile female patients (tubal ligation, hysterectomy or bilateral oophorectomy) may be enrolled.
   3. Agree to abstain from breast feeding during the study participation and for 1 year after the IMP infusion.
9. Male patients must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential for at least 1 year after IMP infusion, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Patient has undergone a prior allogeneic stem cell transplant with either standard or reduced intensity conditioning ≤12 months prior to leukapheresis.
2. Patient has undergone a prior allogeneic stem cell transplant with either standard or reduced intensity conditioning >12 months, and suffers on chronic Graft-versus-Host Disease and/or is on systemic immune-suppressants.
3. Patient with diagnosis of MM

   1. in first relapse following an autologous stem cell transplantation or
   2. in second relapse that subsequently achieves a complete response that is considered being a candidate for an allogeneic stem cell transplantation, unless the patient explicitly denies undergoing an allogeneic stem cell transplantation.
4. Patient has received anti-CD38 and/or anti-SLAMF7 antibodies ≤8 weeks prior to leukapheresis.
5. Ongoing treatment with systemic immune-suppressants (e.g. systemic cyclosporine or systemic steroids at any dose).

   (Note: Physiologic steroid replacement therapy, topical immune-suppressants as e.g. cyclosporine/tacrolimus eye drops and topical steroids are permitted.)
6. Echocardiogram with left ventricular ejection fraction <45%.
7. Inadequate renal function defined by creatinine clearance (CrCl) ≤45 mL/min using Cockcroft-Gault equation.
8. Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN) and total bilirubin >1.5 x ULN (unless due to Gilbert's syndrome and direct bilirubin is ≤1.5 x ULN; unless due to intrahepatic myeloma lesions as demonstrated by MRI or positron emission tomography (PET)/computed tomography (CT) not older than 4 weeks prior to screening).
9. International ratio (INR) or partial thromboplastin time (PTT) >1.5 x ULN, unless on a stable dose of anti-coagulant.
10. Evidence of human immunodeficiency virus (HIV) infection.
11. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV), excluding

    * Patients who are hepatitis B surface antigen negative and HBV viral DNA negative
    * Patients who had hepatitis B but have received an antiviral treatment and show non-detectable viral DNA for 6 months
    * Patients who are seropositive because of hepatitis B virus vaccine
    * Patients with known HBV infection but undetectable HBV viral load and on anti-viral therapy to prevent HBV reactivation.
12. Seropositive for and with active viral infection with hepatitis C virus (HCV), excluding

    - Patients who had hepatitis C but had received an antiviral treatment and show no detectable HCV viral RNA for 6 months.
13. Seropositive for syphilis on treponema pallidum hemagglutination test, excluding

    - Patients with negative treponema pallidum antibody absorption test result
14. Patients with active infection (e.g. asymptomatic and symptomatic severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] infection) or other serious medical or psychiatric disorder on investigators decision.
15. Pregnant or lactating women.
16. Current or previous (within 30 days of enrollment) treatment with another IMP.
17. Known abuse of alcohol, drugs, or medicinal products.
18. Employees of the sponsor, or employees or relatives of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety determination of the treatment with SLAMF7 CAR-T in phase I | through study completion, an average of 2 years
  Type, frequency and severity of AEs in phase I
Determination of the maximum tolerated dose (MTD) and the recommended phase IIa dose of SLAMF7 CAR-T in patients with MM | through study Phase I completion, an average of 2 years
  For the primary endpoint in phase I, the maximum tolerated dose will be determined and recommended for phase IIa.
Safety determination of the treatment with SLAMF7 CAR-T in phases I and IIa | through study completion, an average of 2 years
  Type, frequency and severity of AEs in phase I and IIa
Evaluation of the efficacy, defined as overall response rate (ORR) after treatment with SLAMF7 CAR-T in patients with MM | through study completion, an average of 2 years
  In Phase IIa the efficacy will be evaluated, defined as ORR.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Michael Hudecek, Study Director — University Hospital Wuerzburg
Locations (3):
- Centre Hospitalier Universitaire de Lille, Lille, France
- Early Clinical Trial Unit University Hospital Wuerzburg, Würzburg, Germany
- Clinical Trials Unit, Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- See also: CARAMBA project homepage — https://www.caramba-cart.eu/